CLINICAL TRIAL: NCT03403322
Title: Imediate Effects of Kinesio Tapin in Muscle Activity and Time to Perform Sit to Stand Movement in Children With Cerebral Palsy
Brief Title: Kinesio Taping in Sit to Stand Movement fo Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Santa Catarina (Other)
Responsible Party: Principal Investigator, Adriana Neves Dos Santos, Professor, Reseacher, Universidade Federal de Santa Catarina
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: UFSC-SIGPEX / 201702940
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Cerebral Palsy
Keywords: intervention; children
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person that performed data analysis was blind to all conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First test (Other): All measures were evaluated
  Interventions: Other: Kinesio taping; Other: Without taping
- Second test (Other): All measures were evaluated
  Interventions: Other: Kinesio taping; Other: Without taping

INTERVENTIONS:
Other: Kinesio taping — An experienced physiotherapist placed the base of the Kinesio taping strip, over rectus femoris muscle, 3cm bellow the anterior iliac spine, without tension. From this point, the Kinesio taping was placed up to the upper edge of the patella and stretched to 100% tension. It was, then, bi-sectioned, circled the patella and ended in the tuberosity of the femur, without tension. In order to avoid interference in the electromyography signals, a section was held at Kinesio taping at the point where the electrode was placed.
Other: Without taping — Children performed functional activities without tape

SUMMARY:
Children with Cerebral Palsy (CP) present limited performance of functional activities and activities of daily life. Kinesio taping has been definied as a promising technique for children with CP ans has been extensively used in clinical practice. However, several studies have found a low level of evidence of its effectiveness in healthy individuals. We aim to evaluate the effects of the immediate application of Kinesio taping on the activation of the rectus femoris and anterior tibialis muscles and on the duration of sit-to-stand movement in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with spastic CP
* aged from 5 to 18 years
* Gross Motor Function Classification System levels I and II
* able to understand simple commands
* able to perform the sit-to-stand movement without support

Exclusion Criteria:

* muscle shortening in hamstring, gastrocnemius and hip flexors
* deformities in the lower limbs such as fixed hip and knee flexion that could compromise the sit-to-stand movement
* surgical procedures in the lower limbs and trunk in the previous 12 months
* botulinum toxin injection in the previous 6 months

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Muscle activity | on the day of evaluation
  An electromyography analysis was performed to evaluate the rectus femoris and tibialis anterior activity during the sit-to-stand movement and the five time sit-to-stand test. Electrodes were placed in both lower limbs. Mean root mean square (mRMS) values were used for statistical analysis. Mean root mean square values were normalized by the maximum value of each trial and individual.
Time to perform sit to stand | on the day of evaluation
  Children were seated with hip, knee and ankle flexed at 90°. Both feet were symmetrically positioned shoulder width apart and arms were crossed over the chest. Children should get up from the seat after the verbal command of the evaluator. Children performed the sit-to-stand movement at a speed that simulated the one usually adopted in daily routine
Time to perform five time sit-to-stand test | on the day of evaluation
  Children had to get up and sit down five times as fast as possible. The instructions before starting the test were: "Stand up and sit down as quickly as possible for 5 times. The test will be finished when you return to the seated position the 5th time. Continue the sit-to-stand movement until I ask you to stop. If you try but cannot stand up, just let me know. Ready? go!"

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Santa Catarina, Araranguá, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within one year of study completion